CLINICAL TRIAL: NCT07258160
Title: Evaluation of the Effect of Cordycepin on CD8+ Lymphocytopenia in Patients With Solid Tumors: A Randomized Withdrawal Trial
Brief Title: Evaluation of the Effect of Cordycepin on CD8+ Lymphocytopenia in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JD-LK2025016-A03
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Solid Cancer; Lymphopenia
MeSH Terms: conditions — Lymphopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRaG-1 (Experimental)
  Interventions: Drug: PRaG-1
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRaG-1 — The PRaG-1 cordycepin tablets used in this clinical study were produced by Shengmingyuan Company, which is affiliated with the National Bioprocess Engineering Research Center at Nanjing Tech University. The tablets are oral formulations containing 200 mg of cordycepin per tablet and have obtained national food production approval. The production license number is: SC11332019200201.
  Arms: PRaG-1
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of PRaG-1 in improving CD8+ lymphocytopenia in patients with solid tumors who are tumor-free for more than six months after completing radiotherapy and/or chemotherapy. It will also assess the safety of PRaG-1 Cordycepin in these patients. The main questions it aims to answer are:

Does PRaG-1 increase CD8+ lymphocyte counts by more than 25% in this patient population? Does the effect of PRaG-1 maintain when treatment is discontinued? What are the safety and tolerability profiles of PRaG-1 during and after the treatment period? Participants will receive open-label PRaG-1 (one tablet in the morning and one in the evening) for 14 days, and those who show a response (CD8+ lymphocytes increase by more than 25%) will enter a 14-day randomized withdrawal period, where they will be assigned to continue PRaG-1 or switch to a placebo.

Throughout the study, participants will:

Have their peripheral blood lymphocyte subpopulations tested at baseline and on Days 7 and 14 Undergo safety monitoring for adverse events according to CTCAE 5.0 criteria Provide information on their quality of life during the treatment period Researchers will compare the outcomes of those who continue PRaG-1 to those who receive a placebo to determine if the observed improvement in CD8+ lymphocytes is sustained, which would indicate that the drug is effective in maintaining immune response.

DETAILED DESCRIPTION:
Cordycepin: The PRaG-1 cordycepin tablets used in this clinical study were produced by Shengmingyuan Company, which is affiliated with the National Bioprocess Engineering Research Center at Nanjing Tech University. The tablets are oral formulations containing 200 mg of cordycepin per tablet and have obtained national food production approval. The production license number is: SC11332019200201.

This study is a multicenter, prospective, placebo-controlled, two-stage sequential design, randomized withdrawal trial. Patients with CD8+ lymphocytopenia who have been tumor-free for more than six months following the completion of radiotherapy and/or chemotherapy were screened. All patients first received open-label PRaG-1 at a dose of one tablet in the morning and one tablet in the evening for 14 days. Patients whose CD8+ lymphocytes increased by more than 25% were defined as treatment responders and entered the randomized withdrawal phase. The study population was enrolled in two stages into the open-label phase and then randomized accordingly. The alpha level for the two-stage testing was allocated using the Pocock method (both stages at 0.029). In the first stage, 80 subjects were enrolled in the open-label phase, and 48 of them entered the withdrawal trial. If the first stage met the superiority hypothesis, the trial would terminate; otherwise, it would proceed to the second stage. In the second stage, 47 subjects were enrolled in the open-label phase, and 28 of them entered the withdrawal trial. Data from both stages were combined for the final superiority test. Centralized randomization was used in both stages, with patients assigned in a 1:1 ratio to continue receiving PRaG-1 or to receive a placebo at one tablet in the morning and one tablet in the evening for 14 days. Peripheral blood lymphocyte subpopulations were measured on the day before treatment (baseline), and on Days 7, 14, 21, and 28 of the treatment period. The primary endpoint was the proportion of patients whose CD8+ lymphocytes decreased by more than 25% from baseline after the withdrawal period. Secondary endpoints included lymphocyte dynamics during the entire treatment period and quality of life scores. Safety endpoints included adverse events occurring during treatment and within four weeks after treatment, which were graded according to the CTCAE 5.0 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Participants with solid malignant tumors, with confirmed pathological diagnosis or medical history; they have completed radiotherapy and/or chemotherapy more than six months ago; and peripheral blood CD8+ absolute count (blood drawn before 10:00 AM) below the lower reference limit (LRL);
3. No treatment with immunomodulatory or immunosuppressive agents within the past 2 weeks prior to enrollment;
4. ECOG performance status score of 0-1, with an estimated life expectancy of ≥ 3 months;
5. AST and ALT ≤ 3.0 times the upper limit of normal (ULN) within one week prior to study enrollment; serum creatinine ≤ 2 times ULN;
6. Ability to understand the study and voluntarily provide written informed consent.

Exclusion Criteria:

1. History of uncontrolled epilepsy, central nervous system (CNS) disease, or mental disorders, as determined by the investigator to be clinically significant and potentially interfere with the participant's ability to provide informed consent or comply with medication;
2. Significant (i.e., active) cardiovascular disease, including symptomatic coronary heart disease, congestive heart failure classified as New York Heart Association (NYHA) Class II or worse, or serious arrhythmias requiring pharmacological intervention, or history of myocardial infarction within the past 12 months;
3. Known active serious infections, or in the investigator's opinion, presence of major hematological, renal, metabolic, gastrointestinal, or endocrine dysfunction, or other serious, uncontrolled comorbidities;
4. History of allergy to fungi, or to any of the following components: Cordyceps militaris extract powder, D-mannitol, maltitol, microcrystalline cellulose, or magnesium stearate;
5. History of immunodeficiency, including HIV positive status, or diagnosis with other acquired or congenital immunodeficiencies, or a history of organ transplantation, or immunological disorders requiring long-term oral corticosteroid treatment;
6. Acute gout flare
7. Any other condition deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in CD8+ Proportion of Participants with >25% Decline in CD8+ Lymphocyte During the Withdrawal Period (measured by flow cytometry) | 2 weeks

SECONDARY OUTCOMES:
CD8+ Lymphocyte Response Over Time | 4 weeks
  Peripheral blood CD8+ T cell percentage measured by flow cytometry at baseline, week 1, week 2, and week 4

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China